CLINICAL TRIAL: NCT05757492
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CHS-006, as Monotherapy and in Combination With Toripalimab, in Participants With Advanced Solid Tumors
Brief Title: Study to Evaluate Safety and PK of CHS-006 in Combination With Toripalimab in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated for strategic reasons (not for safety concerns)
Sponsor: Coherus Oncology, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry); Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHS-006-01
Record Dates: First submitted 2023-01-02; First posted 2023-03-07 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor; Non-Small Cell Lung Cancer; Hepatocellular Carcinoma
Keywords: TIGIT inhibitor; PD-1 inhibitor; Advanced Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Hepatocellular | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open-label, multiple-phase, multiple phase study. Participants within the advanced solid tumor dose optimization phase will be assigned to one of two dosing arms. After one CHS-006 dose has been selected from Phase 1, Phase 2 participants will be dosed with that dose in combination with toripalimab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Optimization Phase - Arm A (Active Comparator): Advanced solid tumor participants will receive CHS-006 in combination with toripalimab Q3W
  Interventions: Drug: CHS-006 (anti-TIGIT); Drug: toripalimab (anti-PD-1)
- Dose Optimization Phase - Arm B (Active Comparator): Advanced solid tumor participants will receive CHS-006 in combination with toripalimab Q3W
  Interventions: Drug: CHS-006 (anti-TIGIT); Drug: toripalimab (anti-PD-1)
- Indication-specific Expansion Phase - Cohort 1 NSCLC-NS (Active Comparator): NSCLC-NS participants will receive CHS-006 in combination with toripalimab Q3W
  Interventions: Drug: CHS-006 (anti-TIGIT); Drug: toripalimab (anti-PD-1)
- Indication-specific Expansion Phase - Cohort 2 HCC (Active Comparator): HCC participants will receive CHS-006 in combination with toripalimab Q3W
  Interventions: Drug: CHS-006 (anti-TIGIT); Drug: toripalimab (anti-PD-1)

INTERVENTIONS:
Drug: CHS-006 (anti-TIGIT) — Arm A participants will receive CHS-006 administered via IV Q3W.
  Other Names: JS006
Drug: toripalimab (anti-PD-1) — Arm B participants will receive toripalimab administered via IV Q3W.
  Other Names: CHS-007, TAB001, JS001

SUMMARY:
This phase 1 open-label study will evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of CHS-006 in combination with toripalimab in 2 phases. Phase 1 (Dose Optimization phase) will explore 2 different dose combinations in participants with advanced/metastatic solid tumors (except pancreatic) and Phase 2 (Indication-specific Expansion phase) will use one selected dose in specific tumor types (non-small cell lung cancer-non squamous [NSCLC-NS] and Hepatocellular carcinoma [HCC])

DETAILED DESCRIPTION:
The Dose Optimization phase will enroll participants with advanced/metastatic solid tumors (except pancreatic). Up to 20 participants will be randomized into two dosing arms. Two different primary advanced solid tumors have been selected for investigation of antitumor activity in the Indication-specific Expansion phase. Up to 40 participants will be enrolled into each Indication-specific Expansion phase cohort. All participants in both phases will receive CHS-006 in combination with toripalimab intravenously (IV) every 3 weeks (Q3W).

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥18 years old;
* Histopathologically or cytologically confirmed advanced solid tumor (except pancreatic) with disease progression after at least 1 prior line of standard therapy (Dose Optimization phase);
* Tumor-specific criteria (Indication-specific Expansion phase):
* NSCLC-NS (without sensitizing EGFR/ALK/ROS-1/MET mutations) 2nd line plus (2L+): has received and progressed on at least 1 prior chemotherapy regimen. Prior treatment with both anti-PD-1 therapy and platinum-based chemotherapy either concurrently or sequentially are eligible.
* Hepatocellular carcinoma (HCC) 2L+: has received and progressed on at least 1 prior anticancer regimen. Participants with prior treatment with an anti-PD-1 or PD-L1 agent are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and expected survival ≥12 weeks;
* At least 1 measurable lesion per RECIST v1.1;
* Adequate organ and marrow function

Exclusion Criteria:

* Current or prior use of systemic anticancer therapy, including but not limited to chemotherapy, immunotherapy, biologic therapy, hormone therapy, and targeted therapy, within 28 days prior to the 1st dose of CHS-006;
* NSCLC participants with genomic mutations (e.g., EGFR, ALK, ROS-1, MET, etc.) for which FDA-approved targeted therapies are available or require progression on appropriate prior to enrollment;
* Prior exposure to monoclonal antibodies (mAbs) targeting TIGIT or any of its ligands, including CD155, CD112, or CD113;
* Major surgery within 28 days prior to the 1st dose of CHS-006 or still recovering from prior surgery;
* Symptomatic or untreated central nervous system (CNS) metastases;
* Use of therapeutic immunosuppressive medication within 28 days prior to the 1st planned dose of CHS-006;
* Receipt of live, attenuated vaccination within 30 days prior to the 1st dose of CHS- 006;
* History of active autoimmune disease within the past 2 years, with the following exceptions: vitiligo, alopecia, endocrinopathies controlled by hormone replacement therapy, rheumatoid arthritis and other arthropathies that have not required immunosuppression other than nonsteroidal anti-inflammatory agents, celiac disease controlled by diet, or psoriasis controlled with topical medication;
* Participants with another active solid tumor that has not been curatively treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the number of participants with treatment-emergent adverse events (TEAEs) receiving CHS-006 administered in combination with toripalimab | Day 1 of study treatment through up to 90 days post last dose of study treatment
  Assessed by number of participants with TEAEs assessed by the investigator as per CTCAE v5.0.

SECONDARY OUTCOMES:
Description of the PK profile of CHS-006 in combination with toripalimab | Measured at multiple timepoints from Day 1 of study treatment through up to 90 days post last dose of study treatment
  Assessed by serum concentration of CHS-006 and toripalimab as determined by validated assays
Immunogenicity of CHS-006 and/or toripalimab | Measured at multiple timepoints from Day 1 of study treatment through up to 90 days post last dose of study treatment
  Percentage of participants who develop treatment-emergent antidrug antibodies (ADA) to CHS-006 and/or toripalimab
Objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 assessed by the investigator | Measured at multiple timepoints from Day 1 of study treatment through +/- 7 days at the completion of or premature withdrawal from the study
  Investigator-assessed ORR as per RECIST v1.1
Duration of response (DoR) using RECIST v1.1 assessed by the investigator | Measured at multiple timepoints from Day 1 of study treatment through +/- 7 days at the completion of or premature withdrawal from the study
  Investigator-assessed DoR as per RECIST v1.1
Disease control rate (DCR) using RECIST v1.1 assessed by the investigator | Measured at multiple timepoints from Day 1 of study treatment through +/- 7 days at the completion of or premature withdrawal from the study
  Investigator-assessed DCR as per RECIST v1.1
Time to response (TTR) using RECIST v1.1 assessed by the investigator | Measured at multiple timepoints from Day 1 of study treatment through +/- 7 days at the completion of or premature withdrawal from the study
  Investigator-assessed TTR as per RECIST v1.1
Progression-free survival (PFS) using RECIST v1.1 assessed by the investigator | Measured at multiple timepoints from Day 1 of study treatment through +/- 7 days at the completion of or premature withdrawal from the study
  Investigator-assessed PFS as per RECIST v1.1
Overall survival (OS) using RECIST v1.1 assessed by the investigator | Measured at multiple timepoints from Day 1 of study treatment through +/- 7 days at the completion of or premature withdrawal from the study
  Investigator-assessed PFS as per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Florida Health Cancer Center, Orlando, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Renown Institute for Cancer, Reno, Nevada
  - Gabrail Cancer and Research Center, Canton, Ohio